CLINICAL TRIAL: NCT04404608
Title: Study of the Etiology of Lymphopenia in Covid19 Viral Infection
Brief Title: Etiology of Lymphopenia in Covid19 Infection
Status: Completed | Type: Observational
Sponsor: Dr Medhat Khafagy (Other)
Responsible Party: Sponsor-Investigator, Dr Medhat Khafagy, professor of surgical oncology, Cairo University
Organization: Cairo University (Other)
Other Study IDs: 201920008.2
Record Dates: First submitted 2020-05-23; First posted 2020-05-27 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Lymphopenia
MeSH Terms: conditions — Lymphopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asymptomatic or mild symptoms patients patients: Patients with no or mild symptoms and need no respiratory support.
  Interventions: Diagnostic Test: Complete blood picture, bone marrow aspiration cytology
- Severe symptoms patients: Patients who need admission to ICU because he needs oxygen by nasal canula and needs drugs whether azthromycin or remdesivir according to treatment protocol.
  Interventions: Diagnostic Test: Complete blood picture, bone marrow aspiration cytology
- Critically ill patients: Patients who need artificial ventilation because of many causes and may need plasma from convalescent patients
  Interventions: Diagnostic Test: Complete blood picture, bone marrow aspiration cytology

INTERVENTIONS:
Diagnostic Test: Complete blood picture, bone marrow aspiration cytology — none except the regular routine investigations in such cases

SUMMARY:
Study of the cause of lymphopenia in Covid19 viral infection will be done in 3 cohorts. First cohort will be patients asymptomatic or with mild symptoms. Second cohort will be patients with severe illness and admitted to ICU. Third cohort will be patients critically ill and on artificial ventilation.

DETAILED DESCRIPTION:
Each cohort will include 30 patients. Complete blood count in all patients will be done daily in all patients. Bone marrow aspiration cytology will be done in some selected patients especially those with lymphopenia less than 1000 per cubic mm.

Correlation of the degree of lymphopenia with the status of the patients will be done. Also correlation will be done about the relation of recovery of lymphopenia and status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Any patient admitted with the diagnosis of Covid19 viral infection

Exclusion Criteria:

* Any patient who died within one day of admission

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted with the diagnosis off Covid19 viral infection of all ages and all ethnic backgrounds and agree about the study
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Death or recovery | Up to 24 weeks
  Follow up

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No